CLINICAL TRIAL: NCT02336542
Title: For Tuberculosis (TB) Clinical Auxiliary Diagnosis of Recombinant Mycobacterium Tuberculosis Allergen ESAT6 - CFP10 Dose of Certain Phase IIb Clinical Research
Brief Title: Phase IIb Clinical Study of Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Collaborators: Shanghai Public Health Clinical Center (Other Government); Tianjin Haihe Hospital (Other); Wuhan Institute for Tuberculosis Control (Other); Proswell Medical Corporation (Industry); Air Force Military Medical University, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: LTao-IIb-patient
Record Dates: First submitted 2014-12-24; First posted 2015-01-13 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2015-09

CONDITIONS: Tuberculosis
Keywords: diagnosis of Tuberculosis; ESAT6; CFP10; skin test; diagnostic test
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TB subjects (Experimental): 96 TB subjects are divided into four groups average .24 TB subjects are injected 5μg/ml ESAT6-CFP10 in left arm and TB-PPD in right arm,24 TB subjects are injected 5μg/ml ESAT6-CFP10 in right arm and TB-PPD in left arm,24 TB subjects are injected 10μg/ml ESAT6-CFP10 in left arm and TB-PPD in right arm,24 TB subjects are injected 10μg/ml ESAT6-CFP10 in right arm and TB-PPD in left arm.
  Interventions: Biological: 5μg/ml ESAT6-CFP10 in left arm and TB-PPD in right arm; Biological: 5μg/ml ESAT6-CFP10 in right arm and TB-PPD in left arm; Biological: 10μg/ml ESAT6-CFP10 in left arm and TB-PPD in right arm; Biological: 10μg/ml ESAT6-CFP10 in right arm and TB-PPD in left arm
- non-TB subjects with lung disease (Active Comparator): 96 non-TB subjects with lung disease are divided into four groups average .24 TB subjects are injected 5μg/ml ESAT6-CFP10 in left arm and TB-PPD in right arm,24 TB subjects are injected 5μg/ml ESAT6-CFP10 in right arm and TB-PPD in left arm,24 TB subjects are injected 10μg/ml ESAT6-CFP10 in left arm and TB-PPD in right arm,24 TB subjects are injected 10μg/ml ESAT6-CFP10 in right arm and TB-PPD in left arm.
  Interventions: Biological: 5μg/ml ESAT6-CFP10 in left arm and TB-PPD in right arm; Biological: 5μg/ml ESAT6-CFP10 in right arm and TB-PPD in left arm; Biological: 10μg/ml ESAT6-CFP10 in left arm and TB-PPD in right arm; Biological: 10μg/ml ESAT6-CFP10 in right arm and TB-PPD in left arm

INTERVENTIONS:
Biological: 5μg/ml ESAT6-CFP10 in left arm and TB-PPD in right arm — TB subjects and non-TB subjects with lung disease inject 5μg/ml ESAT6-CFP10 in left arm and TB-PPD in right arm respectively. Two drug must use at the same person and different arm.
Biological: 5μg/ml ESAT6-CFP10 in right arm and TB-PPD in left arm — TB subjects and non-TB subjects with lung disease inject 5μg/ml ESAT6-CFP10 in right arm and TB-PPD in left arm respectively. Two drug must use at the same person and different arm.
Biological: 10μg/ml ESAT6-CFP10 in left arm and TB-PPD in right arm — TB subjects and non-TB subjects with lung disease inject 10μg/ml ESAT6-CFP10 in left arm and TB-PPD in right arm respectively. Two drug must use at the same person and different arm.
Biological: 10μg/ml ESAT6-CFP10 in right arm and TB-PPD in left arm — TB subjects and non-TB subjects with lung disease inject 10μg/ml ESAT6-CFP10 in right arm and TB-PPD in left arm respectively. Two drug must use at the same person and different arm.

SUMMARY:
96 TB subjects and 96 non-TB subjects with lung disease who all meet the standard are divided into different groups through a randomized, blind methods.Every subject inject intradermally ESAT6-CFP10 and TB-PPD in different arms of the same person.Specific γ- IFN(gamma interferon) detection is needed before the injection.Evaluate the sensitivity (positive coincidence rate) ,the specificity (negative coincidence rate) and the coincidence rate of ESAT6-CFP10 in the tuberculosis patients and non-tuberculosis patients with lung diseases, and determine the optimal dose of ESAT6-CFP10 for clinical auxiliary diagnosis of tuberculosis.

DETAILED DESCRIPTION:
Firstly,96 TB(Tuberculosis ) subjects which meet the standard respectively are divided into different groups through a randomized, blind methods.

1. ESAT6-CFP10 （5μg/ml）in left arm；
2. ESAT6-CFP10 （5μg/ml）in right arm；
3. ESAT6-CFP10 （10μg/ml）in left arm；
4. ESAT6-CFP10 （10μg/ml）in right arm； Inject intradermally ESAT6-CFP10 and TB-PPD(tuberculin purified protein derivative ) in different arms of the same subject.For each of the participants in this clinical research, this study uniform that left arm inject a drug(ESAT6-CFP10 or TB - PPD) first, observe 30 min and no no obvious adverse reaction ,then another drug(ESAT6-CFP10 or TB - PPD) inject in right arm. We need draw blood to detect specific γ- IFN before the injection.Observe and record the vital signs (breathing, heart rate, blood pressure and temperature),the skin reaction diameter of injection site (flush and induration) , local reactions (rash, pain, itching and skin mucous membrane) and a variety of adverse events.

Secondly, 96 non-TB subjects with lung disease are divided into different groups and the procedure are as the same as 96 TB subjects above .

Finally,we evaluate the sensitivity (positive coincidence rate) ,the specificity (negative coincidence rate) and the coincidence rate of ESAT6-CFP10 in the TB patients and non-tuberculosis patients with lung diseases,determine the optimal dose of ESAT6-CFP10 for clinical auxiliary diagnosis of tuberculosis,and further evaluate the safety of ESAT6-CFP10 for the clinical auxiliary diagnosis of tuberculosis .

ELIGIBILITY:
Inclusion Criteria of TB (tuberculosis ) subjects:

* Diagnosis TB ;
* 18 to 65 years ;
* Consent and signed informed consent forms(ICF) ;
* Comply with follow-up .

Exclusion Criteria of TB (tuberculosis ) subjects:

* advanced cancer, diabetes,copd in acute episodes, acute/ progressive liver disease or kidney disease, congestive heart failure, etc ;
* Taking part in other clinical or within 3 months involved in any other clinical;
* histories of allergy ;
* in pregnancy or lactation;
* In a mental illness ;
* Any conditions affect the trial evaluation.

Inclusion Criteria of Non-tuberculosis subjects with lung disease :

* Diagnosis non-tuberculosis subjects with lung disease ;
* 18 to 65 years ;
* Consent and signed signed informed consent forms(ICF) ;
* Comply with follow-up .

Exclusion Criteria of Non-tuberculosis subjects with lung disease :

* advanced cancer, diabetes,copd in acute episodes, acute/ progressive liver disease or kidney disease, congestive heart failure, etc ;
* Taking part in other clinical or within 3 months involved in any other clinical;
* histories of allergy;
* in pregnancy or lactation;
* In a mental illness ;
* Any conditions may affect the trial evaluation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
the diameter of induraton or redness within 72 hours after intradermal injection with ESAT6-CFP10 in TB patients | within 72h after injection
  we measure the size 15min,24h,48h,72h after administered intradermally ESAT6-CFP10
the proportion of positive reaction within 72 hours after administered intradermally TB-PPD in TB patient | within 72h after injection
  we measure the size at 15min,24h,48h,72h after administered intradermally TB-PPD
Immune response of of ESAT6-CFP10 from the size of induration OR redness in non-TB patients with lung diseases | within 72h after injection
  we measure the size at 15min,24h,48h,72h after administered intradermally TB-PPD
The proportion of positive reaction after receiving specificity γ-IFN test in TB subjects and non-TB subjects with lung disease | before administered intradermally
the proportion of positive reaction within 72 hours after intradermal injection with TB-PPD in non-TB patients with lung diseases | within 72h after injection
  we measure the size at 15min,24h,48h,72h after administered intradermally TB-PPD

SECONDARY OUTCOMES:
the occurrence of adverse events within 72 hours after injection in TB subjects and non-TB subjects with lung disease | within 72h after injection two drugs
the consistency between ESAT6-CFP10 and TB-PPD in TB subjects and non-TB subjects with lung disease | within 72h after injection
the consistency between ESAT6-CFP10 and γ-IFN in TB subjects and non-TB subjects with lung disease | within 72h after injection
the consistency between TB-PPD and γ-IFN in TB subjects and non-TB subjects with lung disease | within 72h after injection

CONTACTS AND LOCATIONS:
Overall Officials: Shuihua Lu, Bachelor, Principal Investigator — Shanghai Public Health Clinical Center; Qi Wu, Master, Principal Investigator — Tianjin Haihe Hospital; Weihua Wang, Doctor, Principal Investigator — Wuhan Insititute for Tuberculosis Control

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Pinxteren LA, Ravn P, Agger EM, Pollock J, Andersen P. Diagnosis of tuberculosis based on the two specific antigens ESAT-6 and CFP10. Clin Diagn Lab Immunol. 2000 Mar;7(2):155-60. doi: 10.1128/CDLI.7.2.155-160.2000. PMID 10702486
- [Background] Ravn P, Munk ME, Andersen AB, Lundgren B, Lundgren JD, Nielsen LN, Kok-Jensen A, Andersen P, Weldingh K. Prospective evaluation of a whole-blood test using Mycobacterium tuberculosis-specific antigens ESAT-6 and CFP-10 for diagnosis of active tuberculosis. Clin Diagn Lab Immunol. 2005 Apr;12(4):491-6. doi: 10.1128/CDLI.12.4.491-496.2005. PMID 15817755
- [Background] Brusasca PN, Colangeli R, Lyashchenko KP, Zhao X, Vogelstein M, Spencer JS, McMurray DN, Gennaro ML. Immunological characterization of antigens encoded by the RD1 region of the Mycobacterium tuberculosis genome. Scand J Immunol. 2001 Nov;54(5):448-52. doi: 10.1046/j.1365-3083.2001.00975.x. PMID 11696195
- [Background] Weldingh K, Andersen P. ESAT-6/CFP10 skin test predicts disease in M. tuberculosis-infected guinea pigs. PLoS One. 2008 Apr 23;3(4):e1978. doi: 10.1371/journal.pone.0001978. PMID 18431468
- [Background] Aagaard C, Govaerts M, Meikle V, Vallecillo AJ, Gutierrez-Pabello JA, Suarez-Guemes F, McNair J, Cataldi A, Espitia C, Andersen P, Pollock JM. Optimizing antigen cocktails for detection of Mycobacterium bovis in herds with different prevalences of bovine tuberculosis: ESAT6-CFP10 mixture shows optimal sensitivity and specificity. J Clin Microbiol. 2006 Dec;44(12):4326-35. doi: 10.1128/JCM.01184-06. Epub 2006 Sep 27. PMID 17005738
- [Derived] Xu M, Lu W, Li T, Li J, Du W, Wu Q, Liu Q, Yuan B, Lu J, Ding X, Li F, Liu M, Chen B, Pu J, Zhang R, Xi X, Zhou R, Mei Z, Du R, Tao L, Martinez L, Lu S, Wang G, Zhu F. Sensitivity, Specificity, and Safety of a Novel ESAT6-CFP10 Skin Test for Tuberculosis Infection in China: 2 Randomized, Self-Controlled, Parallel-Group Phase 2b Trials. Clin Infect Dis. 2022 Mar 1;74(4):668-677. doi: 10.1093/cid/ciab472. PMID 34021314
- See also: Center for drug evaluation, CFDA ,China — https://wbca.cde.org.cn/wbca/clinmain.do?method=edit&ckmIdCode=8BE5738082A97A9E5471F80B4F814FCF